CLINICAL TRIAL: NCT05561439
Title: Multicenter Retrospective Study of Passive Dosimeter Results for Interventional Cardiologists and Radiologists
Brief Title: Individual Dosimetric Monitoring of Workers During Interventional Radiology and Cardiology Procedures for Cardiologists and Radiologists in France
Acronym: DOSE RPW-CRI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2021-01 /CD-01
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Radiation Exposure

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (16):
- Cardiology: Coronary/Valvular
  Interventions: Other: Dosimetric monitoring
- Cardiology: Rhythmology
  Interventions: Other: Dosimetric monitoring
- Cardiology: Mixed
  Interventions: Other: Dosimetric monitoring
- Radiology: Simple Vascular
  Interventions: Other: Dosimetric monitoring
- Radiology: Complex Vascular
  Interventions: Other: Dosimetric monitoring
- Radiology: Mixed Vascular
  Interventions: Other: Dosimetric monitoring
- Radiology: Simple Osteoarticular
  Interventions: Other: Dosimetric monitoring
- Radiology: Complex Osteoarticular
  Interventions: Other: Dosimetric monitoring
- Radiology: Mixed Osteoarticular
  Interventions: Other: Dosimetric monitoring
- Radiology: Simple Neuroradiology
  Interventions: Other: Dosimetric monitoring
- Radiology: Complex Neuroradiology
  Interventions: Other: Dosimetric monitoring
- Radiology: Mixed Neuroradiology
  Interventions: Other: Dosimetric monitoring
- Radiology: Mixed
  Interventions: Other: Dosimetric monitoring
- Radiology: Simple Oncology
  Interventions: Other: Dosimetric monitoring
- Radiology: Complex Oncology
  Interventions: Other: Dosimetric monitoring
- Radiology: Mixed Oncology
  Interventions: Other: Dosimetric monitoring

INTERVENTIONS:
Other: Dosimetric monitoring — Dosimetric monitoring of workers Information retrieved from passive dosimeters results from the years 2019, 2020 and 2021

SUMMARY:
The objective of this study is to review the results of annual radiation doses received by interventional cardiologists and radiologists in France. The results of this study will allow the improvement of classification of interventional cardiology and radiology activities and procedures to help define radiation dose constraints for occupational exposure, according to the number and types of procedures performed.

The study is based on the hypothesis that some specialties in interventional cardiology (cardiology or rythmology procedures) and in interventional radiology (vascular, neuroradiology, osteoarticular) and some types of procedures present greater exposure risks for interventional cardiologists and radiologists. It is expected that the annual radiation dose limits for workers can be exceeded if good practices for both patient and worker radiation protection are not applied. Also, dosimetry equipment used to detect radiation dose although provided to the workers are not systematically worn by the physician during the procedure . The study is likely to show that for an equivalent speciality and number of procedures per type of act, the correct use of collective and personal radiation protection equipment (préciser) will lower occupational radiation exposure of physician . Similarly, for an equivalent activity and number of procedures per type of act , a trained physician would have a lower occupational exposure than an untrained physician. The physician's radiation exposure should therefore increase with a greater number of procedures per type of procedure performed and as the radiation dose delivered to the patient increase. Finally, there would be a different correlation between patient's radiation dose and physician's exposure depending on specialty, procedures, modality, experience and availability and use of collective and personal radiation protection equipment.

ELIGIBILITY:
Inclusion Criteria:

* Physician performing interventional cardiology or radiology procedures with a fixed C-arm system
* Physician systematically wearing at least one of the following personal dosimeters: whole body, extremities, lens.

Exclusion Criteria:

* Physician who did not perform an interventional procedure during the observation period (2019-2021)
* For the primary endpoint by year, physician with more than 3 months of missing data (more than one 3-month period or more than 3 1-month periods)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in the study will be interventional cardiologists and interventional radiologists exposed to radiation during their interventional procedures performed as part of their activity.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Annual occupational radiation exposure levels for effective dose for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2019
  mSv
Annual occupational radiation exposure levels for effective dose for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2020
  mSv
Annual occupational radiation exposure levels for effective dose for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2021
  mSv
Annual occupational radiation exposure levels for equivalent doses to the skin for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2019
  mSv
Annual occupational radiation exposure levels for equivalent doses to the skin for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2020
  mSv
Annual occupational radiation exposure levels for equivalent doses to the skin for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2021
  mSv
Annual occupational radiation exposure levels for equivalent doses to the lens of the eye for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2019
  mSv
Annual occupational radiation exposure levels for equivalent doses to the lens of the eye for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2020
  mSv
Annual occupational radiation exposure levels for equivalent doses to the lens of the eye for interventional cardiologists and radiologists according to their specialty, activity and type of procedures performed | 2021
  mSv

SECONDARY OUTCOMES:
Availability and frequency of use for each passive dosimeter | 2019
  Yes/no for each passive dosimeter (whole body, extremities, lens) 4 categories: worn systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Availability and frequency of use for each passive dosimeter | 2020
  Yes/no for each passive dosimeter (whole body, extremities, lens) 4 categories: worn systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Availability and frequency of use for each passive dosimeter | 2021
  Yes/no for each passive dosimeter (whole body, extremities, lens) 4 categories: worn systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
High and low radiation protection equipment availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
High and low radiation protection equipment availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
High and low radiation protection equipment availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
High radiation protection alone (ceiling suspension) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
High radiation protection alone (ceiling suspension) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
High radiation protection alone (ceiling suspension) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Low radiation protection alone (windscreen) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Low radiation protection alone (windscreen) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Low radiation protection alone (windscreen) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Radioprotective sterile fields (e.g. RADPAD) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Radioprotective sterile fields (e.g. RADPAD) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Radioprotective sterile fields (e.g. RADPAD) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Arm support systems with a radioprotection (e.g. STARBOARD) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Arm support systems with a radioprotection (e.g. STARBOARD) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Arm support systems with a radioprotection (e.g. STARBOARD) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Lead apron or vests and skirts availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Lead apron or vests and skirts availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Lead apron or vests and skirts availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded collars or thyroid protectors availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded collars or thyroid protectors availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded collars or thyroid protectors availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded sleeves (handle) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019,
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded sleeves (handle) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded sleeves (handle) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded eye protection (glasses, over-glasses or visors) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019, 2020 and 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded eye protection (glasses, over-glasses or visors) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded eye protection (glasses, over-glasses or visors) availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Gloves use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded head caps availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2019
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded head caps availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2020
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Leaded head caps availability and use by interventional physicians according to specialty, activity and type of procedures performed | 2021
  Yes/no; classed as used systematically (100% of the time), often (> 50% of the time), infrequently (<50% of the time) or never (not worn) according to specialty, activity and type of procedures performed
Patient radiation protection training status according to specialty, activity and type of procedures performed | 2019,
  Up-to-date/needs renewing/never completed
Patient radiation protection training status according to specialty, activity and type of procedures performed | 2020
  Up-to-date/needs renewing/never completed
Patient radiation protection training status according to specialty, activity and type of procedures performed | 2021
  Up-to-date/needs renewing/never completed
Worker radiation protection training status according to specialty, activity and type of procedures performed | 2019
  Up-to-date/needs renewing/never completed
Worker radiation protection training status according to specialty, activity and type of procedures performed | 2020
  Up-to-date/needs renewing/never completed
Worker radiation protection training status according to specialty, activity and type of procedures performed | 2021
  Up-to-date/needs renewing/never completed
Physician exposure according to total number of procedures | 2019
  mSv: Information taken from Dosimetry Archiving and Communication System
Physician exposure according to total number of procedures | 2020
  mSv: Information taken from Dosimetry Archiving and Communication System
Physician exposure according to total number of procedures | 2021
  mSv: Information taken from Dosimetry Archiving and Communication System
Physician exposure according to number of procedures by type of specialty | 2019
  mSv: Information taken from Dosimetry Archiving and Communication System
Physician exposure according to number of procedures by type of specialty | 2020
  mSv: Information taken from Dosimetry Archiving and Communication System
Physician exposure according to number of procedures by type of specialty | 2021
  mSv: Information taken from Dosimetry Archiving and Communication System
Physician exposure according to number of procedures by modality | 2219
  mSv: Information taken from Dosimetry Archiving and Communication System
Physician exposure according to number of procedures by modality | 2020
  mSv: Information taken from Dosimetry Archiving and Communication System
Physician exposure according to number of procedures by modality | 2021
  mSv: Information taken from Dosimetry Archiving and Communication System
Relationships between the whole body, extremity and lens radiation exposures and the Dose Area Product patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2019
  Gy.cm²
Relationships between the whole body, extremity and lens radiation exposures and the Dose Area Product patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2020
  Gy.cm²
Relationships between the whole body, extremity and lens radiation exposures and the Dose Area Product patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2021
  Gy.cm²
Relationships between whole body, extremity and lens exposures and the Air Kerma at the interventional reference point patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2019
  mGy
Relationships between whole body, extremity and lens exposures and the Air Kerma at the interventional reference point patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2020
  mGy
Relationships between whole body, extremity and lens exposures and the Air Kerma at the interventional reference point patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2021
  mGy
Relationships between the physician's whole body, extremity and lens exposures and the Dose Length Product patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2019
  mGy.cm
Relationships between the physician's whole body, extremity and lens exposures and the Dose Length Product patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2020
  mGy.cm
Relationships between the physician's whole body, extremity and lens exposures and the Dose Length Product patient dosimetric indicator per physician (dosimetric indicators) according to specialty, activity and type of procedures performed | 2021
  mGy.cm

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Duverger, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France